CLINICAL TRIAL: NCT02912364
Title: Double-Blind, Randomized, Two Period Crossover Comparison of the Cognitive and Behavioral Effects of Eslicarbazepine Acetate and Carbamazepine in Healthy Adults
Brief Title: Comparison of the Cognitive and Behavioral Effects of Eslicarbazepine Acetate and Carbamazepine in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Kimford Jay Meador, Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 34098
Record Dates: First submitted 2016-09-14; First posted 2016-09-23 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-04

CONDITIONS: Epilepsy
Keywords: Eslicarbazepine; Carbamazepine; cognition
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine; eslicarbazepine acetate; Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eslicarbazepine (Experimental): Randomized to eslicarbazepine 800mg po bid in crossover design.
  Interventions: Drug: Eslicarbazepine
- Carbamazepine (Experimental): Randomized to carbamazepine 400mg po bid in crossover design.
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Eslicarbazepine — Healthy adults will be titrated onto Eslicarbazepine Acetate (800mg daily) . After four weeks maintenance they will be tapered off and enter washout period, then crossed over to 2nd drug.
  Other Names: Aptiom
  Arms: Eslicarbazepine
Drug: Carbamazepine — Healthy adults will be titrated onto Carbamazepine (400 mg bid). After four weeks maintenance they will be tapered off and enter washout period, then crossed over to 2nd drug.
  Other Names: Tegretol
  Arms: Carbamazepine

SUMMARY:
Double-blind, randomized, two period crossover comparison of the cognitive and behavioral effects of Eslicarbazepine acetate and Carbamazepine in healthy volunteers.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, two period crossover design. The study consists of 6 visits over a 21 week period. Forty six (46) normal healthy subjects will be treated with both Eslicarbazepine acetate (ESL, 800 mg/day) and Carbamazepine (CBZ, 800mg/day) for 6 weeks and 3 days each (maintenance 4 weeks and taper 3 days). Each antiepileptic drug (AED) treatment period will be followed by a four day taper and washout period off AED for the remainder of the month. Cognitive and behavioral testing along with safety testing will be conducted at pretreatment baseline, the end of each randomization AED maintenance period, and after the final washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between the ages of 18 and 55 years old.
2. Male or female

Exclusion Criteria:

1. Presence of clinically significant cardiovascular, endocrine, hematopoietic, hepatic, neurologic, psychiatric, or renal disease or pregnancy.
2. Presence or history of drug or alcohol abuse.
3. The use of concomitant medications, which are known to affect ESL or Carbamazepine or the use of any concomitant medications that may alter cognitive function (see Section VII.E for a partial list).
4. Use of oral contraceptive hormones or other medications that could be affected by ESL or Carbamazepine.
5. Prior adverse reaction to or prior hypersensitivity to either study medication or to related compounds.
6. Prior participation in studies involving anticonvulsant medications.
7. Subjects who have received any investigational drug within the previous thirty days.
8. Subjects with IQ < 70 as determined by the Peabody Picture Vocabulary Test.
9. Presence of HLA B*1502 in subjects of Asian descent; this will be obtained at screening in subjects of Asian descent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimford Meador, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Eslicarbazepine, Then Carbamazepine: Healthy adults will be titrated onto Eslicarbazepine Acetate (800mg once daily). After four weeks maintenance they will be tapered off and enter washout period, then crossed over to receive Carbamazepine, 400mg twice daily.
- Carbamazepine, Then Eslicarbazepine: Healthy adults will be titrated onto Carbamazepine (400mg twice daily). After four weeks maintenance they will be tapered off and enter washout period, then crossed over to Eslicarbazepine Acetate, 800mg daily.
Period: Treatment 1
Arm/Group | Eslicarbazepine, Then Carbamazepine | Carbamazepine, Then Eslicarbazepine
Started | 23 | 23
Received Intervention | 18 | 18
Completed | 13 | 11
Not Completed | 10 | 12
Period: Washout Period
Arm/Group | Eslicarbazepine, Then Carbamazepine | Carbamazepine, Then Eslicarbazepine
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0
Period: Treatment 2
Arm/Group | Eslicarbazepine, Then Carbamazepine | Carbamazepine, Then Eslicarbazepine
Started | 13 | 11
Received Intervention | 12 | 11
Completed | 12 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants who received either Eslicarbazepine Acetate (800mg once daily), or Carbamazepine, 400mg twice daily.
Arm/Group | All Participants
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3
  Asian | 13
  Hispanic/Latino | 6
  White/Caucasian | 24
Education Level [Mean (Standard Deviation); unit: years] — Education level is reported as the average number of years spent in school.
  years | 15.0 (1.9)
IQ Estimate [Mean (Standard Deviation); unit: units on a scale] — IQ scores are generally interpreted as follows
  * Over 140 - Genius or near genius
  * 120 - 140 - Very superior intelligence
  * 110 - 119 - Superior intelligence
  * 90 - 109 - Normal or average intelligence
  * 80 - 89 - Dullness
  * 70 - 79 - Borderline deficiency
  * Under 70 - Definite feeble-mindedness
  units on a scale | 98.6 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: Overall Composite Z Score of Neuropsychological Battery as a Measure of Direct Comparison of the 2 Antiepileptic Drugs.
Description: Z score of cognitive tests at end of each 6-week drug treatment period for each intervention (i.e., Eslicarbazepine and Carbamazepine). The Z-score indicates the number of standard deviations away from a reference population. A Z-score of 0 is equal to the mean. Negative numbers indicate poor cognitive performance compared to the mean and positive numbers represent higher cognitive performance compared to the mean.
Time Frame: At the end of each 6-week drug treatment period.
Population: Participants who completed the protocol are included in the analysis. That is, participants who completed both treatment arms (completed treatment 2 in the participant flow) are included in the analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Eslicarbazepine: Eslicarbazepine Acetate (800mg once daily).
- Carbamazepine: Carbamazepine (400mg twice daily).
Arm/Group | Eslicarbazepine | Carbamazepine
Number analyzed (Participants) | 12 | 11
Z-score | .001 (.50) | -.23 (.61)
Statistical Analysis 1: Comparison: Eslicarbazepine vs Carbamazepine; Test type: Other; p < .001, t-test, 2 sided; degrees of freedom = 22; Mean Difference (Final Values) = .23, 95% CI 2-sided [.13 to .34]

2. Secondary Outcome: Overall Z-score for Executive Function.
Description: Executive function consists of a composite of measures from the computerized cognitive tests. The Z-score indicates the number of standard deviations away from a reference population. A Z-score of 0 is equal to the mean. Negative numbers indicate poor cognitive performance compared to the mean and positive numbers represent higher cognitive performance compared to the mean.
Time Frame: At the end of each 6-week drug treatment period.
Population: Participants who completed the protocol are included in the analysis. That is, participants who completed both treatment arms (Eslicarbazepine and Carbamazepine) are included in the analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Eslicarbazepine | Carbamazepine
Number analyzed (Participants) | 12 | 11
Z-score | .22 (.53) | -.32 (.76)
Statistical Analysis 1: Comparison: Eslicarbazepine vs Carbamazepine; Test type: Other; p < .001, t-test, 2 sided; Degrees of freedom = 22; Mean Difference (Final Values) = .54, 95% CI 2-sided [.30 to .79]

3. Secondary Outcome: MCG Paragraph Recall Scores.
Description: Participants were read a paragraph and were asked to recall content immediately following and twenty minutes after hearing the reading. MCG = Medical College of Georgia.
  Assessments were performed prior to treatment (non-drug condition average) and at the end of each treatment period. Score range: 0 - 60, higher scores indicate better memory function.
Time Frame: Prior to treatment (non-drug condition average) and at the end of each six-week treatment period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Non-drug Condition Average: Average of scores prior to treatment 1 and treatment 2.
Arm/Group | Non-drug Condition Average | Eslicarbazepine | Carbamazepine
Number analyzed (Participants) | 23 | 12 | 11
units on a scale
  Immediate Recall | 34 (17) | 33 (12) | 31 (15)
  Delayed Recall | 33 (18) | 31 (13) | 30 (16)

4. Secondary Outcome: Dual Task Percent of Time in Box.
Description: Participants were asked to use their computer mouse to keep the cursor inside a moving box on the computer screen while simultaneously responding with a button press when a number on the screen exceeded a certain value.
  Assessments were performed prior to treatment (non-drug condition average) and at the end of each treatment period.
Time Frame: Prior to treatment (non-drug condition average) and at the end of each six-week treatment period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time in box
Arm/Group | Non-drug Condition Average | Eslicarbazepine | Carbamazepine
Number analyzed (Participants) | 23 | 12 | 11
percentage of time in box | 62 (33) | 62 (33) | 60 (34)

5. Secondary Outcome: Profile of Mood States (POMS) Score.
Description: Participants were asked to rate the extent to which they feel a variety of emotions/feelings. The overall score is presented.
  Assessments were performed prior to treatment (non-drug condition average) and at the end of each treatment period. Score range: -32 to 200. Lower scores correspond to better mood state.
Time Frame: Prior to treatment (non-drug condition average) and at the end of each six-week treatment period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-drug Condition Average | Eslicarbazepine | Carbamazepine
Number analyzed (Participants) | 23 | 12 | 11
units on a scale | 8 (25) | 11 (29) | 15 (32)

ADVERSE EVENTS:
Time Frame: Up to 21 weeks
Arm/Group | Eslicarbazepine | Carbamazepine
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 12/29 | 21/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eslicarbazepine (N=29) | Carbamazepine (N=30)
Agitation (Nervous system disorders) | 0 | 1
Altered pitch perception (pitch seemed lower) (Nervous system disorders) | 0 | 1
Clouded vision (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Coordination/balance problems (Nervous system disorders) | 0 | 1
Difficulty naming objects (Nervous system disorders) | 0 | 1
Disorientation (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 4
Drowsiness (Nervous system disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 10 | 9
Grogginess (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 3
Headache (mild) (Nervous system disorders) | 0 | 1
Hot Flashes (Nervous system disorders) | 0 | 1
Hunger (General disorders) | 1 | 0
Lightheadedness (Nervous system disorders) | 0 | 2
Loopy Feeling (Nervous system disorders) | 0 | 1
Loss of taste (Nervous system disorders) | 0 | 1
Memory problems (Nervous system disorders) | 1 | 1
Minor muscle twitch in hands (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Sleepiness (Nervous system disorders) | 0 | 1
Twitching (Nervous system disorders) | 0 | 1
Upset stomach (Gastrointestinal disorders) | 0 | 1
Visual Illusions (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT02912364/Prot_SAP_000.pdf